CLINICAL TRIAL: NCT01668446
Title: Effect of Adding Sildenafil to Protocol of Endometrial Preparation in Outcome of Frozen-thawed Embryo Transfer Cycles
Acronym: sildenafil
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: farzaneh hojjat (Other)
Collaborators: Razieh dehghani firouzabadi (Unknown); Robab davar (Unknown)
Responsible Party: Sponsor-Investigator, farzaneh hojjat, Farzaneh hojjat MD, Shahid Sadoughi University of Medical Sciences and Health Services
Organization: Shahid Sadoughi University of Medical Sciences and Health Services (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: radvin123; rad123 (Other: Shahid Sadoughi University of Medical Science); rad123 (Other: Shahid Sadoughi University of Medical Science, Bouali Ave. Safaieh, Yazd,Iran.)
Record Dates: First submitted 2012-06-24; First posted 2012-08-20 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Endometrial Preparation; Frozen Embryo Transfer
Keywords: Sildenafil; Endometrial thickness; Frozen embryo transfer; ultrasonographic endometrial thickness; endometrial pattern; Implantation rate; chemical pregnancy rate
MeSH Terms: interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sildenafil (Experimental): One of two group to prepare the endometrium give estradiol by step up method with menstruation.
  From first to fourth day of menstrual cycle, estradiol valerat tablet 2 mg daily From Fifth to eighth day of menstrual cycle, estradiol valerat tablet 4 mg daily From Ninth to twelfth day of menstrual , estradiol valerat tablet 6 mg daily The second group in addition to the above treatment protocol from First day of cycle until day of starting progesterone will be given sildenafil tablets(50 mg) daily.
  Interventions: Drug: Sildenafil
- Sildenafil and estradiol valerat (Experimental): One of two group to prepare the endometrium give estradiol by step up method with menstruation.
  From first to fourth day of menstrual cycle, estradiol valerat tablet 2 mg daily From Fifth to eighth day of menstrual cycle, estradiol valerat tablet 4 mg daily From Ninth to twelfth day of menstrual , estradiol valerat tablet 6 mg daily The second group in addition to the above treatment protocol from First day of cycle until day of starting progesterone will be given sildenafil tablets(50 mg) daily.
  Interventions: Drug: Sildenafil; Drug: estradiol valerat

INTERVENTIONS:
Drug: Sildenafil — sildenafil tablets(50 mg) daily
Drug: estradiol valerat
  Arms: Sildenafil and estradiol valerat

SUMMARY:
The target of this study was an estimate the result of sildenafil on ultrasonographic endometrial thickness, endometrial pattern investigation estrogen level on the day of progesterone administration, Implantation rate and chemical pregnancy rate in frozen embryo transfer cycles .

ELIGIBILITY:
Inclusion Criteria:

* women > 40 years old,
* history of endocrine disease
* Hysteroscopic surgery
* cardiovascular, renal and liver disease
* hypotension( blood pressure < 90/50)
* history of stroke or myocardial infarction
* use of alcohol or substance

Exclusion Criteria:

A total of 80 patients with antecedent of poor endometrial response and had frozen embryo included in this study all women must to be < 40 years old,

* no history of endocrine disease,
* no Hysteroscopic surgery, had a high quality embryos no cardiovascular,
* renal and liver disease and
* no hypotension (blood pressure < 90/50) or
* history of stroke or myocardial infarction and
* don't use of alcohol or substance Patients with these conditions enter this study and based on randomized tables are divided in two groups.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2009-09; Primary Completion 2009-09 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
estimate the result of sildenafil on ultrasonographic endometrial thickness | between 2009-2011 (up to 2 years)
  Assays:
  Day 13 of menstrual cycle endometrial thickness estimated with Transvaginal ultrasonographic(arranged in a series every other day), evaluations were performed by a single investigator, If the endometrial thickness is more than 8mm progesterone injected 100 mg intramuscular and Estrogen, progesterone and lh measured in blood sample then after three days embryo transferred.

SECONDARY OUTCOMES:
estimate the result of sildenafil on Implantation rate and chemical pregnancy rate in frozen embryo transfer cycles . | between 2009-2011 (up to 2 years)
  Implantation rate was higher in sildenafil Group but not significant chemical pregnancy rates were higher in sildenafil Group but not significant.

CONTACTS AND LOCATIONS:
Overall Officials: farzaneh hojjat, MD, Principal Investigator — Department of Obstetrics and Gynecology, Research and Clinical Center for Infertility, Shahid Sadoughi University of Medical Science, Bouali Ave. Safaieh, Yazd,Iran.
Locations (1):
- Farzaneh Hojjat, Yazd, Iran